CLINICAL TRIAL: NCT00232089
Title: Assessment of Efficacy and Safety of Tegaserod Treatment and Placebo in Women With Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919D2302
Record Dates: First submitted 2005-09-08; First posted 2005-10-04 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Dyspepsia
Keywords: Dyspepsia, gastrointestinal, tegaserod
MeSH Terms: conditions — Dyspepsia | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study is being done to evaluate the safety, tolerability and satisfactory relief of dyspepsia symptoms in females excluding those with predominant stomach pain. Tegaserod will be evaluated at 6mg twice daily and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 18 years and older
* Self-reported presence of persistent or recurrent adverse digestive symptoms consistent with dyspepsia; for at least 12 weeks, not necessarily consecutive, during the previous 12 months.

Exclusion Criteria:

* Abnormal esophago-gastro-duodenoscopy (EGD) endoscopy findings such as any esophageal mucosal break, gastric erosions, gastric ulcers and/or duodenal ulcers/erosions on an EDG exam performed with 12 weeks prior to baseline.
* Current or history of erosive esophagitis confirmed by EGD
* Heartburn occurring 3 or more days a week.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 1296
Dates: Start 2004-05; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Over 6 weeks of treatment assessment of percent of days with satisfactory relief of dyspepsia and/or average severity score in (average of postprandial fullness early satiety and bloating)

SECONDARY OUTCOMES:
Weekly assessment of satisfactory relief of dyspepsia.
Daily assessment of percentage of patients responding on average severity score.
For each week assessment of average daily severity score.
Percentage of days with satisfactory relief of dyspepsia during each week.
Weekly global assessment of change in dyspepsia condition.
Weekly assessment of individual symptoms score of postprandial fullness early satiety, bloating, abdominal pain, nausea and vomiting.
Quality of life at end of treatment compared to baseline.
Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — East Hanover NJ
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Vakil N, Laine L, Talley NJ, Zakko SF, Tack J, Chey WD, Kralstein J, Earnest DL, Ligozio G, Cohard-Radice M. Tegaserod treatment for dysmotility-like functional dyspepsia: results of two randomized, controlled trials. Am J Gastroenterol. 2008 Aug;103(8):1906-19. doi: 10.1111/j.1572-0241.2008.01953.x. Epub 2008 Jul 4. PMID 18616658